CLINICAL TRIAL: NCT07299422
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of SHR-2173 Injection in Patients With Systemic Lupus Erythematosus
Brief Title: A Study of SHR-2173 in Participants With Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-2173-202
Record Dates: First submitted 2025-11-28; First posted 2025-12-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-2173 Injection Group (Experimental)
  Interventions: Drug: SHR-2173 Injection
- SHR-2173 Injection Placebo Group (Placebo Comparator)
  Interventions: Drug: SHR-2173 Injection Placebo

INTERVENTIONS:
Drug: SHR-2173 Injection — SHR-2173 injection in different doses.
  Arms: SHR-2173 Injection Group
Drug: SHR-2173 Injection Placebo — SHR-2173 injection placebo.
  Arms: SHR-2173 Injection Placebo Group

SUMMARY:
This study is a randomized, double-blind, multi-center, placebo-controlled Phase II clinical trial to evaluate the efficacy and safety of SHR-2173 in adult participants with active Systemic Lupus Erythematosus (SLE), including a 4-week screening period, a 24-week core treatment period, a 24-week maintenance treatment period, and a 12-week safety follow-up period. Approximately 245 SLE patients will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18 through 65 years (including boundary value)at the time of screening.
2. The Body Mass Index (BMI) ≥18 kg/m ² at the time of screening.
3. Diagnosed with SLE for at least 6 months prior to screening.
4. ANA≥1:80, or anti-dsDNA antibodies and/or anti-Sm antibodies above the upper limit of the normal range as determined by a central laboratory at the time of screening.
5. High disease activity at screening and at baseline.
6. Currently receiving at least one or more of the following standard therapies for SLE at stable doses: oral corticosteroids (OCS), antimalarial drugs, and conventional immunosuppressants.
7. Participants thoroughly understand the content, process and possible adverse reactions before the trial, and voluntarily sign the written informed Consent Form (ICF).
8. Female subjects with fertility or male participants whose partners are women of childbearing age must avoid donating sperm/eggs from the date of signing the ICF until 12 weeks after the last study medication, and agree to take contraceptive measures as specified in the protocol.

Exclusion Criteria:

1. The presence of any of the following medical histories or comorbidities: a) Severe lupus-related kidney disease and/or kidney damage; b) Active neuropsychiatric SLE occurred 6 months prior to screening; c) Autoimmune, inflammatory or joint diseases other than SLE and LN that may interfere with the interpretation of the test results or clinical assessment, including but not limited to rheumatoid arthritis, overlap syndrome, psoriasis/psoriatic arthritis, eczema, inflammatory bowel disease, and any other vasculitis; d) There was catastrophic or severe antiphospholipid syndrome within 12 months prior to screening; e) Have a history of progressive multifocal leukoencephalopathy (PML); f) Have a history of organ transplantation.
2. Use any of the following medications /treatments or participate in a clinical trial: a) Previously received gene therapy such as CAR-T or T-cell Engager (TCE) ; b) Received anti-CD20 monoclonal antibody within 6 months and other B-cell or plasma cell depletion treatments within 6 to 12 months prior to randomization; c) Received biologic therapy targeting BAFF, APRIL or interferon receptor within 12 weeks prior to randomization; d) Received Alkylating agents within 12 weeks prior to randomization; e) Received any other biological agents for the treatment of SLE within 12 weeks prior to randomization; f) Received inhibitors of Janus kinase (JAK), Bruton tyrosine kinase (BTK), or tyrosine kinase 2 (TYK2) within 12 weeks prior to randomization; g) Received intra-articular, intramuscular or intravenous corticosteroid for SLE within 4 weeks prior to randomization; h) Received a live/attenuated live vaccine within 4 weeks prior to randomization or planned to receive it during the trial period.
3. The presence of the following tumor risks or accompanied by other poorly controlled serious or chronic diseases: a) Suffering from malignant tumors or having a history of malignant tumors; b) Accompanying other poorly controlled serious or chronic diseases during or at the time of screening, including but not limited to endocrine diseases, cardiovascular diseases, neurological/mental disorders, kidney diseases, severe digestive system diseases, severe respiratory system diseases, neurological diseases, and other serious liver, gallbladder, metabolic or lymphatic system diseases, etc.
4. Infection-related medical history and examinations: a) Herpes zoster infection meets one of the following conditions: 1) A history of systemic herpes zoster, such as disseminated herpes zoster, herpetic encephalitis or ocular herpes zoster involving the retina; 2) Recurrent herpes zoster that has occurred twice or more within two years; 3) The herpes zoster infection has not completely subsided within 12 weeks before screening; b) Tuberculosis (TB) or occult tuberculosis infection; c) A history of primary immunodeficiency, splenectomy, and any potential conditions that make participants susceptible to infection; d) A history of repeated infections requiring hospitalization and intravenous antibiotics; e) Hospitalization and/or intravenous anti-infective treatment were required within 8 weeks prior to randomization, or any infection that required oral anti-infective treatment within 2 weeks prior to randomization; f) Positive test results for any of the following: hepatitis B surface antigen (HBsAg), hepatitis C virus antibody, Treponema pallidum antibody or human immunodeficiency virus (HIV); If the test result is negative for HBsAg but positive for hepatitis B core antibody (HBcAb), regardless of whether the hepatitis B surface antibody (HBsAb) is positive or negative, HBV-DNA testing is required to determine the situation: if HBV-DNA is positive, participants should be excluded. Participants can be included if HBV-DNA is negative.
5. General situation: a) Pregnant or lactating women; b) Having a history of alcohol abuse or illegal drug abuse within one year prior to screening; c) Individuals with allergic constitutions, or those known to be intolerant or allergic to any component of the investigational drug; d) Participants who have undergone major surgeries within the 3 months prior to screening, or those who plan to undergo major surgeries during the trial period; e) Investigators determine that there are circumstances that affect the safety and efficacy evaluation of the investigational drug, or other circumstances not appropriate for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants achieving Systemic Lupus Erythematosus Responder Index-4 (SRI-4) at Week 24. | At Week 24.

SECONDARY OUTCOMES:
The proportion of participants achieving SRI-4. | Up to Week 48.
The proportion of participants achieving British Isles Lupus Assessment Group(BILAG) based Composite Lupus Assessment (BICLA). | Up to Week 48.
The proportion of participants with a ≥ 4-point decrease from baseline in SLE Disease Activity Index 2000 (SLEDAI-2K). | Up to Week 48.
The proportion of participants achieving SRI-4 on low-dose corticosteroids in the protocol. | Up to Week 48.
The proportion of participants with a daily prednisone (or equivalent) dose of ≤ 7.5 mg (limited to those with baseline corticosteroids > 7.5 mg/day). | Up to Week 48.
Change from baseline in Patient's Global Assessment(PGA). | Up to Week 48.
The proportion of participants achieving Lupus Low Disease Activity State (LLDAS) in the protocol. | Up to Week 48.
The proportion of participants achieving Definitions of Remission In SLE (DORIS) in the protocol. | Up to Week 48.
Change from baseline in the level of anti-dsDNA antibody. | Up to Week 48.
Change from baseline in the level of complement (C3, C4). | Up to Week 48.
Change from baseline in the level of CD19+B cells. | Up to Week 48.
Change from baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) in the protocol. | Up to Week 48.
Changes from baseline in SLE-Specific Quality-Of-Life (SLEQOL) in the protocol. | Up to Week 48.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided